CLINICAL TRIAL: NCT07364409
Title: Restoration of Spermatogenesis by Autologous Grafting of Cryopreserved Testis Tissue From Men With Non-Obstructive Azoospermia and Healthy Men With Proven Fertility
Brief Title: Autologous Transplantation of Human Cryopreserved Testis Tissue
Acronym: ReSTORE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Collaborators: University of Copenhagen (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Elena von Rohden, MD, PhD fellow, Herlev and Gentofte Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-24039098; 2096-00027B (Other Grant/Funding Number: Independent Research Fund Denmark (DFF)); P-2024-17175 (Registry Identifier: Privacy (Capital Region of Denmark's research registry))
Record Dates: First submitted 2025-12-13; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-10

CONDITIONS: Cancer; Hematologic Diseases; Infertility, Male; Azoospermia, Nonobstructive
MeSH Terms: conditions — Neoplasms; Hematologic Diseases; Infertility, Male; Azoospermia, Nonobstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous Transplantation of Testis Tissue (Experimental): Autologous transplantation of testis tissue under the scrotal skin
  Interventions: Procedure: Autologous Transplantation of Testis Tissue

INTERVENTIONS:
Procedure: Autologous Transplantation of Testis Tissue — Autologous transplantation of testis tissue under the scrotal skin

SUMMARY:
For pre-pubertal boys undergoing gonadotoxic therapies, freezing immature testicular tissue (ITT) containing spermatogonial stem cells (SSCs) is currently the only option to potentially preserve future fertility. This experimental clinical study aims to provide proof-of-concept that frozen-thawed, ectopically autotransplanted adult human testicular tissue can support spermatogenesis in healthy adult men.

DETAILED DESCRIPTION:
As of 2025, more than 3,000 pre-pubertal boys worldwide have cryopreserved immature testicular tissue, and the number of centers offering this fertility preservation option prior to gonadotoxic therapies continues to grow. The most advanced strategy for future fertility restoration is the ectopic autologous transplantation of frozen-thawed ITT, allowing the tissue to mature, initiate spermatogenesis, and ultimately provide sperm for assisted fertility treatments.

However, the absence of human data and the preservation of ITT samples for later clinical trials have so far hindered clinical translation. To address this knowledge gap, the investigators will conduct a proof-of-concept study involving five healthy adult participants with normal spermatogenesis who have naturally conceived children and do not desire additional biological offspring.

Participants will be recruited from the Department of Urology, Copenhagen University Hospital, Herlev and Gentofte Hospital. During elective hydrocele or spermatocele surgery, testicular biopsies will be collected and cryopreserved. At a later stage, the frozen-thawed tissue fragments will be autotransplanted ectopically beneath the scrotal skin. Over a six-month period, participants will undergo regular follow-up. At the end of this period, the transplanted tissue will be retrieved and evaluated for the presence of sperm. If spermatozoa are identified, their genetic stability will also be assessed. This study will generate essential data on the safety, feasibility, and functional potential of using cryopreserved human testicular tissue for fertility restoration, thereby supporting the advancement of this approach toward clinical implementation.

ELIGIBILITY:
Men referred to the Department of Urology at Herlev and Gentofte Hospital for the treatment of hydrocele or spermatocele were provided with detailed information about the study and invited to participate. Written study information was distributed, and a mandatory reflection period of at least 24 hours was observed prior to obtaining consent.

Inclusion Criteria:

* Age ≥ 40 years
* Scheduled for an elective hydrocele or spermatocele surgery
* Willing to have a testis biopsy taken during the planned surgery
* At least one biological child, unassisted spontaneous conception
* No current or future fertility wishes
* Written informed consent for the participation in this study

Exclusion Criteria:

* Treatment with testosterone substitution
* Bleeding disorders that render surgery too high a risk
* Other contraindications to surgery
* Unable to give informed consent
* Language difficulties that could compromise the informed consent or quality of examination

Min Age: 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-12-17 (Actual); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Sperm retrieval | Sperm retrieved yes/no at 6 months post transplantation
  The primary outcome of interest is the retrieval of viable sperm by testicular sperm extraction (TESE) from the transplanted testicular tissue

SECONDARY OUTCOMES:
Genetic Stability of retrieved Spermatozoa | Assessed in sperm retrieved 6 months after transplantation
  If spermatozoa are retrieved, the genome will be sequenced to assess gentic stability of sperm retrieved after autotransplantation of frozen-thawed testicular tissue
Histology of engrafted testicular Tissue | Tissue retrieved 6 months after transplantation
  The autotransplanted and retrieved testicular tissue and potentially sperm will be assessed and characterized histopathologically
Safety of subcutaneous Transplantation | From obtaining the testicular biopsy until full healing from the procedure for retrieving the transplanted tissue, up to 3 months after tissue retrieval
  Complications at any point during the study period will be recorded and classified according to Clavien-Dindo

CONTACTS AND LOCATIONS:
Overall Officials: Elena von Rohden, MD, Principal Investigator — Department of Urology, Copenhagen University Hospital - Herlev and Gentofte
Locations (1):
- Copenhagen University Hospital - Herlev and Gentofte, Herlev, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No
Risk of re-identification of individual participants due to small sample size